CLINICAL TRIAL: NCT00040066
Title: Development of Human Laboratory Study Model of Cocaine Relapse Prevention
Brief Title: Development of Human Laboratory Study Model of Cocaine Relapse Prevention. - 1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-CTO-0013-1
Record Dates: First submitted 2002-06-18; First posted 2002-06-18 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2004-09

CONDITIONS: Cocaine-Related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Cocaine

INTERVENTIONS:
Procedure: Cocaine (IV)

SUMMARY:
The purpose of this study is to assess the development of human laboratory study model of cocaine relapse prevention.

DETAILED DESCRIPTION:
The primary objective of this study will be to develop experimental procedures and parameters demonstrating arousal and craving responses to cocaine-related environmental cues as a model for future testing of the relapse prevention medication treatment of cocaine addiction.

ELIGIBILITY:
Inclusion Criteria:

* Cocaine dependent, non treatment seeking individuals

Exclusion Criteria:

Please contact site directly for details.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32
Dates: Start 2002-05; Study Completion 2003-08

PRIMARY OUTCOMES:
Cocaine craving
Cocaine related high

CONTACTS AND LOCATIONS:
Overall Officials: John Roache, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (2):
- United States (2):
  - UCLA Integrated Substance Abuse Program, Los Angeles, California
  - University of Texas Health Science Center, San Antonio, Texas